CLINICAL TRIAL: NCT03385915
Title: Nationwide Finnish Registry of Transcatheter and Surgical Aortic Valve Replacement for Aortic Valve Stenosis: FinnValve Registry
Brief Title: Finnish Registry of Transcatheter and Surgical Aortic Valve Replacement for Aortic Valve Stenosis: FinnValve Registry
Acronym: FinnValve
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Fausto Biancari, Professor, Turku University Hospital
Other Study IDs: T309/2017
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter aortic valve replacement; Transcatheter aortic valve implantation; TAVI; TAVR; Aortic valve replacement; Surgical aortic valve replacement; Sutureless
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAVI cohort: Patients who underwent transcatheter aortic valve implantation for aortic valve stenosis
  Interventions: Procedure: Aortic valve replacement
- SAVR cohort: Patients who underwentsurgical aortic valve replacement for aortic valve stenosis
  Interventions: Procedure: Aortic valve replacement

INTERVENTIONS:
Procedure: Aortic valve replacement — Transcatheter or surgical aortic valve replacement for severe aortic valve stenosis

SUMMARY:
The FinnValve investigators planned a nationwide registry to investigate the early and late outcome of transcatheter aortic valve implantation (TAVI) compared to surgical aortic valve replacement (SAVR) in patients with aortic valve stenosis performed from 2008 to 2017 at five Finnish University Hospitals. Data will be collected in a dedicated electronic case report form.

DETAILED DESCRIPTION:
Rationale of the study Uncertainty regarding the potential benefits of transcatheter aortic valve implantation (TAVI) compared to surgical aortic valve replacement (SAVR) in patients with aortic valve stenosis (AS) requires well-designed studies with long-term data on the outcome of these patients. A Finnish nationwide registry would allow complementing of the knowledge gained from randomized trials by providing data on the outcome of a more inclusive patient population, within a Health Care System that reflects the actual clinical practice in Scandinavia. In fact, the internal validity attained in randomized trials is often achieved at the expense of uncertainty about generalizability, especially since the populations enrolled in such studies may differ in significant ways from those seen in practice.

The choice among different surgical aortic valve prostheses is based on solid data with 20-year follow-up, which have shown significant risk of structural valve deterioration of bioprosthesis on the second decade after implantation. However, much less is known about the structural durability of TAVI prostheses beyond 3 years of follow-up. This nationwide registry would provide data on the durability of surgical bioprostheses as well as second and third generation TAVI prostheses at 7 years . Continuous follow-up of these patients will allow monitoring of the durability of these prostheses on the long run.

Furthermore, the introduction of TAVI prompted a rapid development of minimally invasive surgical techniques and rapid deployment surgical bioprostheses in order to reduce the risk of early adverse events after SAVR. However, it is unclear whether these advances have a real clinical benefit on the early and late outcome of patients undergoing SAVR.

Patients and Methods

Patients operated on for AS at each Finnish University Hospitals from January 2008 to September 2017 will included in to this registry. The following inclusion and exclusion criteria will be considered:

Inclusion criteria:

* Patients aged >18 years
* Primary aortic valve procedure with a bioprosthesis for AS with or without associated regurgitation.
* TAVI and SAVR with or without associated coronary revascularization
* TAVI and SAVR for AS after any prior major cardiac surgery with exception of any maze procedure and/or closure of the left atrial appendage.

Exclusion criteria:

* Patients who underwent any prior SAVR or TAVI
* Patients undergoing concomitant procedures on the mitral valve, tricuspid valve or the ascending aorta.
* Patients operated on for aortic valve endocarditis
* Patients operated for isolated aortic valve regurgitation.

Definition criteria for baseline and operative variables as well as early and late outcomes will be according to the Valve Academic Research Consortium (VARC) 2 guidelines (Kappetein et al. Eur J Cardiothorac Surg 2012;42:S45-60). Prosthetic valve structural deterioration and failure will be reported according to the last specific guidelines on this topic (Capodanno et al. Eur J Cardiothorac Surg. 2017;52:408-417). However, because of the lack of complete echocardiographic follow-up in these patients, valve structural valve deterioration will be classified only according to the definition criteria of severe hemodynamic structural valve deterioration of these guidelines.

The late events of interest are all-cause mortality, stroke, myocardial infarction, myocardial revascularization, structural deterioration, non-structural valve dysfunction, repeated procedures on the aortic valve and implantation of permanent pace-maker. Data on these late events will be collected at each participating center. These will be further checked and implemented for patients residing outside the catchment areas by interrogation of the Finnish National Health Institute for Health and Welfare database as well as Statistics Finland database.

Planned studies

The following is a tentatile of study projects which will be accomplished from the FinnValve registry:

1. Late outcome of TAVI versus SAVR in intermediate risk patients
2. Late outcome of TAVI versus SAVR in low risk patients
3. Late outcome of TAVI and SAVR in high risk patients
4. Futility of TAVI (3-month analysis)
5. Mini- versus full-sternotomy SAVR
6. Perceval sutureless bioprosthesis: 5-year outcome
7. Late outcome of sutureless versus conventional stented bioprosthesis in isolated SAVR
8. Late outcome of sutureless SAVR versus transfemoral TAVI in low- and intermediate risk patients
9. Early and late outcome of TAVI versus SAVR in patients with recent acute heart failure
10. Early and late outcome of TAVI versus SAVR in bicuspid AS
11. Early and late outcome of TAVI versus SAVR in obese patients (BMI >29) at low- and intermediate risk
12. Early and late outcome of isolated TAVI versus TAVI plus percutaneous coronary intervention (PCI) in patients with coronary artery disease
13. Early and late outcome of TAVI plus PCI versus SAVR plus coornary artery bypass grafting (CABG)
14. Prognostic impact of Syntax score on the early and late outcome after TAVI
15. Early and late outcome of TAVI vs. SAVR in patients with prior CABG
16. Early and late outcome of second versus third generation TAVI prostheses
17. Early and late outcome of transfemoral versus transaortic TAVI
18. Early and late outcome of trans-subclavian artery versus trans-aortic TAVI
19. Early and late outcome of sutureless versus conventional stented bioprosthesis in SAVR plus CABG
20. Early and late outcome of Trifecta versus Perimount bioprosthesis in isolated SAVR
21. Thromboembolic events after TAVI and SAVR
22. Early and late outcome of TAVI in nonagenarians
23. Prognostic impact of permanent pace-maker implantation on the early and late outcome after TAVI and SAVR
24. Prognostic impact of mild paravalvular leakage on the late outcome after SAVR
25. Impact of preoperative atrial fibrillation on the late outcome of TAVI
26. Impact of preoperative atrial fibrillation on the late outcome of SAVR
27. Early and late outcome of TAVI vs. SAVR in patients aged 85 years or older

Publications of results and PhD studies

The results of these studies will be published in international, peer-reviewed journals in the fields of cardiology and cardiac surgery. Furthermore, data from this registry will be available for several doctoral study projects. At this stage, a proposal for PhD studies has been submitted by:

1. Marko Virtanen, MD (Tampere University Hospital);
2. Pasi Maaranen, MD (Tampere University Hospital)
3. Maina Jalava, MD (Turku University Hospital);
4. Tuomas Ahvenvaara (Oulu University Hospital);
5. Teemu Laakso (Helsinki University Hospital).

Time schedule of data collection, checking and analysis

* December 2017: start of data collection
* End of April 2018: deadline for data collection
* End of May 2018: data checking
* June 2018-December 2019: analyses and writing of the planned studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent transcatheter (TAVI) or surgical aortic valve replacement (SAVR) for severe aortic valve stenosis
* Patients aged >18 years
* Primary aortic valve procedure with a bioprosthesis for AS with or without associated regurgitation.
* TAVI and SAVR with or without associated coronary revascularization
* TAVI and SAVR for AS after any prior major cardiac surgery with exception of any maze procedure and/or closure of the left atrial appendage.

Exclusion Criteria:

* Patients who underwent any prior SAVR or TAVI
* Patients undergoing concomitant procedures on the mitral valve, tricuspid valve or the ascending aorta.
* Patients operated on for aortic valve endocarditis
* Patients operated for isolated aortic valve regurgitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent transcatheter (TAVI) or surgical aortic valve replacement (SAVR) for severe aortic valve stenosis at five Finnish University Hospitals from January 2008 to September 2017
Sampling Method: Non-Probability Sample
Enrollment: 6463 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Death | From the index procedure till the end of the follow-up period (December 2017)
  All-cause death

SECONDARY OUTCOMES:
Atrial fibrillation | During the index hospital stay, an average of 7 days
  Any episode of atrial fibrillation
Permanent pace-maker implantation | From the index procedure till the end of the follow-up period (December 2017)
  Permanent pace-maker implantation
Stroke | From the index procedure till the end of the follow-up period (December 2017)
  Stroke
Infection | During the index hospital stay, an average of 7 days
  Deep sternal wound infection/mediastinitis, vascular access site infection, pneumonia, sepsis
Acute kidney injury | During the index hospital stay, an average of 7 days
  Postoperative acute kidney injury according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Bleeding | During the index hospital stay, an average of 7 days
  Minor, major, life-threatening or disabling bleeding according to the VARC 2 definition criteria
Reoperation for bleeding | During the index hospital stay, an average of 7 days
  Reoperation for bleeding
Postoperative intra-aortic balloon pump | During the index hospital stay, an average of 7 days
  Postoperative use of intra-aortic balloon pump
Venoarterial extracorporeal oxygenation | During the index hospital stay, an average of 7 days
  Postoperative use of venoarterial extracorporeal oxygenation
Intensive care unit stay | During the index hospital stay, an average of 7 days
  Length of stay in the intensive care unit
Structural valve deterioration | From the index procedure till the end of the follow-up period (December 2017)
  * Mean transprosthetic gradient ≥40 mmHg
  * Mean transprosthetic gradient ≥20 mmHg change from baseline
  * Severe intraprosthetic regurgitation, new or worsening (>2+/4+) from baseline
Prosthesis thrombosis | From the index procedure till the end of the follow-up period (December 2017)
  Any thrombus attached to or near an implanted valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment
Prosthesis endocarditis | From the index procedure till the end of the follow-up period (December 2017)
  Prosthesis endocarditis requiring medical or surgical treatment
Repeat procedure | From the index procedure till the end of the follow-up period (December 2017)
  Repeat procedure on the aortic valve
Myocardial infarction | From discharge after the index procedure till the end of the follow-up period (December 2017)
  Myocardial infarction occurring after discharge after the index procedure
Coronary revascularization | From the index procedure till the end of the follow-up period (December 2017)
  Coronary revascularization after discharge after the index procedure
Paravalvular regurgitation | During the index hospital stay, an average of 7 days
  Paravalvular regurgitation immediately after the index procedure
TAVI/SAVR prosthesis migration | During the index hospital stay, an average of 7 days
  TAVI/SAVR prosthesis migration
Annulus rupture | During the index hospital stay, an average of 7 days
  Rupture of the aortic annulus
Coronary artery ostium occlusion | During the index hospital stay, an average of 7 days
  Coronary artery ostium occlusion during the index procedure
Ventricular septal perforation | During the index hospital stay, an average of 7 days
  Ventricular septal perforation during the index procedure
Mitral valve apparatus damage or dysfunction | During the index hospital stay, an average of 7 days
  Mitral valve apparatus damage or dysfunction during the index procedure
Tamponade | During the index hospital stay, an average of 7 days
  Pericardial tamponade during or immediately after the index procedure
Vascular injury | During the index hospital stay, an average of 7 days
  Vascular injury during the index procedure
Injury of the left ventricle wall | During the index hospital stay, an average of 7 days
  Injury of the left ventricle wall during the index procedure
Need of emergency cardiac surgery | During the index hospital stay, an average of 7 days
  Need of emergency cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center, Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Jalava MP, Savontaus M, Ahvenvaara T, Laakso T, Virtanen M, Niemela M, Tauriainen T, Maaranen P, Husso A, Kinnunen E, Dahlbacka S, Jaakkola J, Rosato S, D'Errigo P, Laine M, Makikallio T, Raivio P, Eskola M, Valtola A, Juvonen T, Biancari F, Airaksinen J, Anttila V. Transcatheter and surgical aortic valve replacement in patients with left ventricular dysfunction. J Cardiothorac Surg. 2022 Dec 18;17(1):322. doi: 10.1186/s13019-022-02061-9. PMID 36529781
- [Derived] Husso A, Airaksinen J, Juvonen T, Laine M, Dahlbacka S, Virtanen M, Niemela M, Makikallio T, Savontaus M, Eskola M, Raivio P, Valtola A, Biancari F. Transcatheter and surgical aortic valve replacement in patients with bicuspid aortic valve. Clin Res Cardiol. 2021 Mar;110(3):429-439. doi: 10.1007/s00392-020-01761-3. Epub 2020 Oct 24. PMID 33099681
- [Derived] Laakso T, Laine M, Moriyama N, Dahlbacka S, Airaksinen J, Virtanen M, Husso A, Tauriainen T, Niemela M, Makikallio T, Valtola A, Eskola M, Juvonen T, Biancari F, Raivio P. Impact of paravalvular regurgitation on the mid-term outcome after transcatheter and surgical aortic valve replacement. Eur J Cardiothorac Surg. 2020 Dec 1;58(6):1145-1152. doi: 10.1093/ejcts/ezaa254. PMID 33057657
- [Derived] Virtanen MPO, Eskola M, Savontaus M, Juvonen T, Niemela M, Laakso T, Husso A, Jalava MP, Tauriainen T, Ahvenvaara T, Maaranen P, Kinnunen EM, Dahlbacka S, Laine M, Makikallio T, Valtola A, Raivio P, Rosato S, D'Errigo P, Vento A, Airaksinen J, Biancari F. Mid-term outcomes of Sapien 3 versus Perimount Magna Ease for treatment of severe aortic stenosis. J Cardiothorac Surg. 2020 Jun 29;15(1):157. doi: 10.1186/s13019-020-01203-1. PMID 32600369
- [Derived] Biancari F, Dahlbacka S, Juvonen T, Virtanen MPO, Maaranen P, Jaakkola J, Laakso T, Niemela M, Tauriainen T, Vento A, Husso A, Savontaus M, Laine M, Makikallio T, Raivio P, Eskola M, Rosato S, Anttila V, Airaksinen J, Valtola A. Favorable outcome of cancer patients undergoing transcatheter aortic valve replacement. Int J Cardiol. 2020 Sep 15;315:86-89. doi: 10.1016/j.ijcard.2020.03.038. Epub 2020 Mar 18. PMID 32216975
- [Derived] Virtanen MPO, Airaksinen J, Niemela M, Laakso T, Husso A, Jalava MP, Tauriainen T, Maaranen P, Kinnunen EM, Dahlbacka S, Rosato S, Savontaus M, Juvonen T, Laine M, Makikallio T, Valtola A, Raivio P, Eskola M, Biancari F. Comparison of Survival of Transfemoral Transcatheter Aortic Valve Implantation Versus Surgical Aortic Valve Replacement for Aortic Stenosis in Low-Risk Patients Without Coronary Artery Disease. Am J Cardiol. 2020 Feb 15;125(4):589-596. doi: 10.1016/j.amjcard.2019.11.002. Epub 2019 Nov 19. PMID 31831151
- [Derived] Moriyama N, Laakso T, Biancari F, Raivio P, Jalava MP, Jaakkola J, Dahlbacka S, Kinnunen EM, Juvonen T, Husso A, Niemela M, Ahvenvaara T, Tauriainen T, Virtanen M, Maaranen P, Eskola M, Rosato S, Makikallio T, Savontaus M, Valtola A, Anttila V, Airaksinen J, Laine M. Prosthetic valve endocarditis after transcatheter or surgical aortic valve replacement with a bioprosthesis: results from the FinnValve Registry. EuroIntervention. 2019 Aug 9;15(6):e500-e507. doi: 10.4244/EIJ-D-19-00247. PMID 31113766
- [Derived] Makikallio T, Jalava MP, Husso A, Virtanen M, Laakso T, Ahvenvaara T, Tauriainen T, Maaranen P, Kinnunen EM, Dahlbacka S, Jaakkola J, Airaksinen J, Anttila V, Savontaus M, Laine M, Juvonen T, Valtola A, Raivio P, Eskola M, Niemela M, Biancari F. Ten-year experience with transcatheter and surgical aortic valve replacement in Finland. Ann Med. 2019 May-Jun;51(3-4):270-279. doi: 10.1080/07853890.2019.1614657. Epub 2019 May 21. PMID 31112060